CLINICAL TRIAL: NCT05099471
Title: Efficacy of Venetoclax in Combination With Rituximab in Waldenström's Macroglobulinemia
Acronym: VIWA-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christian Buske (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Zentrum für Klinische Studien Ulm (Other); AbbVie (Industry); Pfizer (Industry); University of Ulm (Other); University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor-Investigator, Christian Buske, Prof. Dr., University of Ulm
Organization: University of Ulm (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIWA-1
Record Dates: First submitted 2021-10-04; First posted 2021-10-29 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Waldenstrom Macroglobulinemia; Treatment Naive
Keywords: Hematology; Oncology; Venetoclax; Rituximab; DRC; Lymphoma; NHL; indolent; monoclonal IgM
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Neoplasms; Lymphoma | interventions — venetoclax; Rituximab; Dexamethasone; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venetoclax / Rituximab (Experimental): Cycle 1 (28-days cycle) Stepwise dose escalation of Venetoclax in all patients with a target dose of xy mg/d QD PO.
  Day 1-7: Venetoclax xy mg/d QD PO Day 8-14: Venetoclax xy mg/d QD PO Day 15-28: Venetoclax xy mg/d QD PO
  Cycle 2-12:
  Day 1: Rituximab 375 mg/m2 IV Day 1-28: Venetoclax xy mg/d QD PO
  Interventions: Drug: Venetoclax; Rituximab
- Dexamethasone / Rituximab / Cyclophosphamide (Active Comparator): Cycle 1-6:
  Day 1: Dexamethasone 20 mg PO Day 1: Rituximab 375 mg/m2 IV Day 1-5: Cyclophosphamide 100 mg/m2 BID PO
  Interventions: Drug: DRC

INTERVENTIONS:
Drug: Venetoclax; Rituximab — Combination of venetoclax and rituximab
  Other Names: Venetoclax / Rituximab
  Arms: Venetoclax / Rituximab
Drug: DRC — Combination of Dexamethasone / Rituximab / Cyclophosphamide
  Other Names: Dexamethasone / Rituximab / Cyclophosphamide
  Arms: Dexamethasone / Rituximab / Cyclophosphamide

SUMMARY:
In Waldenström's macroglobulinemia (WM) chemotherapy induces only low CR/VGPR rates and response duration is limited. In addition, WM patients are often elderly, partly not tolerating chemotherapy related toxicities. Thus, innovative approaches are needed which combine excellent activity and tolerability in WM. Chemotherapy-free approaches are highly attractive for this patient group. Based on its high activity and favorable toxicity profile in indolent B-NHL such as CLL, Venetoclax was approved for the treatment of this diseases by the FDA and the European Medicines Agency (EMA). First data in relapsed/refractory WM have documented high activity and low toxicity of Venetoclax also in WM, including patients with prior Ibrutinib treatment or patients carrying CXCR4 mutations. Ibrutinib itself has high activity and a relatively low toxicity profile in WM, but has also major disadvantages: the main disadvantage is the need to apply this drug continuously. Furthermore, Ibrutinib efficacy depends largely on the genotype with a substantial drop in major responses and PFS in the presence of CXCR4 mutations and non-mutated MYD88. In particular the need of continuous treatment for Ibrutinib has prevented that Ibrutinib has become the standard of care outcompeting conventional Rituximab/chemotherapy. This is reflected in current guidelines such as the NCCN and the ESMO guidelines, which still see immunochemotherapy as a backbone of treatment, largely because of the advantage of a timely fixed application. Data in CLL in the relapsed as well as in the first line setting have convincingly shown that in contrast to Ibrutinib Venetoclax is highly efficient also when used in a timely defined application scheme over 12 months in combination with the anti-CD20 antibody Rituximab. Data documented deep responses including molecular responses and a highly significant advantage over immunochemotherapy in large international Phase III trials, changing the standard of care in this disease.

Based on this the hypothesis is that timely fixed application of the combination of Venetoclax and Rituximab induces significantly superior treatment outcomes compared to chemotherapy and Rituximab (DRC) in patients with treatment naïve WM, regardless of the genotype. A first indication for this assumption in the proposed trial will allow the performance of confirmatory phase 3 trials that might change the standard of care in WM.

DETAILED DESCRIPTION:
In Waldenström's macroglobulinemia (WM) chemotherapy induces only low CR/VGPR rates and response duration is limited. In addition, WM patients are often elderly, partly not tolerating chemotherapy related toxicities. Thus, innovative approaches are needed which combine excellent activity and tolerability in WM. Chemotherapy-free approaches are highly attractive for this patient group. Based on its high activity and favorable toxicity profile in indolent B-NHL such as CLL, Venetoclax was approved for the treatment of this diseases by the FDA and the European Medicines Agency (EMA). First data in relapsed/refractory WM have documented high activity and low toxicity of Venetoclax also in WM, including patients with prior Ibrutinib treatment or patients carrying CXCR4 mutations. Ibrutinib itself has high activity and a relatively low toxicity profile in WM, but has also major disadvantages: the main disadvantage is the need to apply this drug continuously. Furthermore, Ibrutinib efficacy depends largely on the genotype with a substantial drop in major responses and PFS in the presence of CXCR4 mutations and non-mutated MYD88. In particular the need of continuous treatment for Ibrutinib has prevented that Ibrutinib has become the standard of care outcompeting conventional Rituximab/chemotherapy. This is reflected in current guidelines such as the NCCN and the ESMO guidelines, which still see immunochemotherapy as a backbone of treatment, largely because of the advantage of a timely fixed application. Data in CLL in the relapsed as well as in the first line setting have convincingly shown that in contrast to Ibrutinib Venetoclax is highly efficient also when used in a timely defined application scheme over 12 months in combination with the anti-CD20 antibody Rituximab. Data documented deep responses including molecular responses and a highly significant advantage over immunochemotherapy in large international Phase III trials, changing the standard of care in this disease.

Based on this the hypothesis is that timely fixed application of the combination of Venetoclax and Rituximab induces significantly superior treatment outcomes compared to chemotherapy and Rituximab (DRC) in patients with treatment naïve WM, regardless of the genotype. A first indication for this assumption in the proposed trial will allow the performance of confirmatory phase 3 trials that might change the standard of care in WM.

This study is an International phase II explorative, multicenter, open label, and randomized trial.

The study will consist of an open labeled, stratified 1:1 randomization between Arm A and Arm B for de novo WM patients in need of treatment (phase II). Stratification factors are MYD88 and CXCR4 status (positive vs. negative). A stratified central block randomization will be used. The central randomization service will be used to avoid predictability of the treatment arm.

The primary goal of this study is to explore the efficacy of Venetoclax plus Rituximab versus Dexamethasone/Cyclophosphamide/Rituximab in the treatment of de novo WM patients (Arm A vs. Arm B).

80 patients are planned to be recruited for this study at approcimately 30 sites in Germany, Greece and France.

ELIGIBILITY:
Inclusion Criteria:

* Proven clinicopathological diagnosis of WM as defined by consensus panel one of the Second International Workshop on WM (IWWM). Histopathology has to be perfomed before randomization but within the last 4 months before start of treatment. In addition, pathological specimens have to be sent to the national pathological reference center prior to randomization for the determination of the mutational status of MYD88 and CXCR4 prior to randomization if the mutational status hasn't been determined before. Pathological reference center must confirm the diagnosis of WM.
* De novo WM independent of the genotype.
* Patients must have at least one of the following criteria to start study treatment as partly defined by consensus panel criteria from the Seventh IWWM and ESMO Guideline:

  * Recurrent fever, night sweats, weight loss, fatigue (at least one of them).
  * Hyperviscosity.
  * Lymphadenopathy which is either symptomatic or bulky (≥ 5 cm in maximum diameter).
  * Symptomatic hepatomegaly and / or splenomegaly.
  * Symptomatic organomegaly and / or organ or tissue infiltration.
  * Peripheral neuropathy due to WM.
  * Symptomatic cryoglobulinemia.
  * Symptomatic Cold agglutinin anemia.
  * Autoimmune hemolytic anemia and/or thrombocytopenia.
  * Nephropathy related to WM.
  * Amyloidosis related to WM.
  * Hemoglobin ≤ 10 g/dL (patients should not have received red blood cells transfusions for at least 7 days prior to obtaining the screening hemoglobin).
  * Platelet count < 100 x 109/L (caused by bone marrow [BM] infiltration of the lymphoma).
  * Serum monoclonal protein > 5 g/dL, even with no overt clinical symptoms.
  * IgM serum concentration ≥ 6 g/dL.
  * and other WM associated relevant symptoms
* Subject must be ≥ 18 years of age.
* Life expectancy > 3 months.
* World Health Organization (WHO) / ECOG performance status ≤ 2.
* Left ventricular ejection fraction ≥ 40% as assessed by transthoracic echocardiogram (TTE).
* Baseline platelet count ≥ 50x109/L, absolute neutrophil count ≥ 0.75x109/L (if not due to BM infiltration by the lymphoma).

  . Adequate hepatic function per local laboratory reference range as follows:
  * Aspartate transaminase (AST) and alanine transaminase (ALT) < 3.0 x ULN.
  * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin).
* Subject must have adequate renal function as demonstrated by a creatinine clearance ≥ 30 mL/min; calculated by the Cockcroft Gault formula or measured by 24 hours urine collection.
* Women of childbearing potential (WCBP), i.e. fertile, following menarche and until becoming postmenopausal must have negative results for pregnancy test and must agree to use a highly effective method of birth control for the duration of the therapy up to 12 months after end of therapy
* Men must agree not to father a child for the duration of therapy and 12 months after and must agree to advice their female partner to use a highly effective method of birth control. Males must refrain from sperm donation for the duration of treatment and at least 12 months after the last dose of study medication.
* Each patient must voluntarily date and sign an informed consent form in the native language of the patient indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study. Patients must be willing and able to adhere to the prohibitions and restrictions specified in this protocol.
* Affiliation to a social security scheme (relevant for France only).

Exclusion Criteria:

* Serious medical or psychiatric illness (especially undergoing treatment) likely to interfere with participation in this clinical study.
* Subject is known to be positive for HIV.
* Active severe infection
* Congenital or acquired severe immunodeficiency not attributed to lymphoma (clinical appearance: recurrent infections, necessity of immunoglobulin substitution therapy, patients after transplantation)
* Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * Uncontrolled systemic infection (viral, bacterial or fungal).
  * Chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate
* inadequate pulmonary function as demonstrated by DLCO ≤ 65% or FEV1 ≤ 65%.
* Creatinine clearance ≥ 30 mL/min to < 45 ml/min
* Uncontrolled diabetes mellitus (as indicated by metabolic derangements and / or severe diabetes mellitus related uncontrolled organ complications).
* Uncontrolled hypertension.
* Cardiac history of CHF requiring treatment or Ejection Fraction ≤ 50% or chronic stable angina.
* Unstable angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months prior to start therapy.
* Clinically significant cardiac arrhythmia that is symptomatic or requires treatment, or asymptomatic sustained ventricular tachycardia.
* Subject has a cardiovascular disability status of New York Heart Association Class > 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea, or anginal pain.
* History of stroke or intracranial haemorrhage within 6 months prior start of treatment
* Known pericardial disease.
* Known interstitial lung disease.
* Infiltrative pulmonary disease, known pulmonary hypertension.
* Prior history of malignancies unless the subject has been free of the disease for ≥ 3 years. Exceptions include the following:

  * Basal cell carcinoma of the skin,
  * Squamous cell carcinoma of the skin,
  * Carcinoma in situ of the cervix,
  * Carcinoma in situ of the breast,
  * Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b).
* Known cirrhosis (meeting child-pugh stage C).
* Chemotherapy with approved or investigational anticancer therapeutic within 21 days prior to start of therapy
* Glucocorticoid therapy within 14 days prior to therapy that exceeds a cumulative dose of 160 mg of dexamethasone or equivalent dose of other corticosteroids given for anti-neoplastic intent.
* Treatment with any of the following within 7 days prior to the first dose of study drug:

  * moderate or strong cytochrome P450 3A (CYP3A) inhibitors (such as fluconazole, ketoconazole, and clarithromycin).
  * moderate or strong CYP3A inducers (such as rifampin, carbamazepine, phenytoin, St. John's wort).
* Contraindication to the active substances or any of the other excipients of the Investigational Medicinal Products as well as to any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs.
* Vaccination with live attenuated vaccines within 4 weeks prior to start of therapy.
* History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or sponsor, if consulted, would pose a risk to subject safely or interfere with the study evaluation, procedures or completion.
* Women who are pregnant as well as women who are breast-feeding and do not consent to discontinue breast-feeding.
* Participation in another clinical trial within four weeks before start of therapy in this study.
* No consent for registration, storage and processing of the individual disease-characteristics.
* Administration or consumption of any of the following within 3 days prior to the first dose of study drug:

  * grapefruit or grapefruit products.
  * Seville oranges (including marmalade containing Seville oranges).
  * star fruit.
* Person of legal age who is incapable of comprehending the nature, significance and implications of the clinical trial and of determining his/her will in the light of these facts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2033-03 (Estimated)

PRIMARY OUTCOMES:
Rate of CR / VGPR | 12 months
  CR / VGPR 12 months after randomization

SECONDARY OUTCOMES:
Interim reponse | 12 months
  response at C4D1; C7D1 (arm A) / 28 days after C6D1 (arm B); C10D1 (arm A) / post treatment staging 1 (arm B) (categories: CR, VGPR, PR, MR, SD, PD, death)
Response rate | 12 months
  response rates (CR, VGPR, PR, MR, SD, PD, death)
Best response | 24 months
  Best response is determined in the time interval from start of treatment up to 24 months (categories: CR, VGPR, PR, MR, SD, PD, death).
Time to first overall response | 24 months
  Time to first overall response is defined as the time from randomization to first overall response (MR, PR, VGPR or CR) within 24 months from start of treatment.
Time to first major response | 24 months
  Time to first major response is defined as the time from randomization to first major response the patient achieves (CR, VGPR, PR) within 24 months from start of treatment.
Event free survival (EFS) | 12 months
  EFS is defined as the date of randomization to the first event of death from any cause or progression or stop of treatment due to toxicity or add-on of new anti-cancer therapy.
Response duration (RD) | 12 months
  Remission duration will be calculated in patients with overall response (CR, VGPR, PR, MR) from the first date of response to the date of progression, relapse or death from any cause.
Progression Free Survival (PFS) | 6 years
  PFS will be calculated from the date of randomization to the following events: the date of progression and the date of death if it occurred earlier.
Lymphoma specific survival (LSS) | 6 years
  Lymphoma specific survival is defined as the period from randomization to death from lymphoma or lymphoma related cause (e.g. infections, bleeding, amyloid caused organ failure).
Overall survival (OS) | 6 years
  Overall survival is defined as the period from randomization to death from any cause. Patients who have not died until the time of the analysis will be censored at their last contact date.
Safety of participants including number of adverse events according to NCI-CTCAE v5.0, SAEs, laboratory parameters, ECG and vital signs. | 12 months
  Adverse events according to NCI-CTCAE version 5.0, SAEs, laboratory parameters (hematology, serum chemistry, b2-microglobulin, coagulation, urine analysis, quantitative immunoglobulins, serum free light chain, cold agglutinin test, serum protein electrophoresis, serum immunofixation, Anti-HIV, HBV, HCV), 12-lead ECG (including PR-, QT- and QTc interval), vital signs (heart rate, blood pressure and temperature)
Quality of life assessed by FACT-Lym questionnaire | 12 months
  Quality of Life will be assessed by the FACT-Lym questionnaire which is a scoring instrument to measure the management of chronic illness in lymphoma patients. A higher score indicates a better quality of life
Comparison of response rates between CXCR4 mutated and CXCR4 wildtype patients | 12 months
  Response rates of CXCR4 mutated and CXCR4 wildtype patients will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Buske, Prof. Dr., Principal Investigator — University Hospital Ulm Department of Internal Medicine III
Locations (11):
- Germany (10):
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Klinikverbund Allgaeu gGmbH, Kempten
  - Universitaetsklinikum Schleswig-Holstein AöR, Kiel
  - Gemeinschaftsklinikum Mittelrhein gGmbH, Koblenz
  - Dr. Vehling-Kaiser MVZ GmbH, Landshut
  - Kliniken Maria Hilf GmbH Moenchengladbach, Mönchengladbach
  - Haematologie und Onkologie Muenchen-Pasing MVZ GmbH, München
  - Universitaet Muenster, Münster
  - University Hospital Ulm, Ulm
- Alexandra Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Buske C, Dimopoulos MA, Morel P. Reply to S. Sarosiek et al. J Clin Oncol. 2023 Aug 20;41(24):4060-4061. doi: 10.1200/JCO.23.00877. Epub 2023 Jun 22. No abstract available. PMID 37348018